CLINICAL TRIAL: NCT00072852
Title: Phase II Trial of Irinotecan in Patients With Advanced Metastatic Breast Cancer Who Have Experienced Failure of an Anthracycline, a Taxane, and Capecitabine
Brief Title: Irinotecan in Patients With Advanced Metastatic Breast Cancer Who Have Experienced Failure of an Anthracycline, a Taxane, and Capecitabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPTAPO-0047-146; A5961023
Record Dates: First submitted 2003-11-11; First posted 2003-11-13 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Irinotecan

INTERVENTIONS:
Drug: Irinotecan

SUMMARY:
The purpose of this phase II, randomized, open-label clinical trial is to study 2 schedules of single-agent Irinotecan in women with metastatic breast cancer who have experienced failure of prior therapy with an anthracycline, a taxane, and capecitabine. Patients will receive Irinotecan capsules either once each day for 5 days, or once a day for 14 days in 3 week cycles.

ELIGIBILITY:
Inclusion Criteria:

* Women with diagnosis of primary adenocarcinoma of the breast
* Presence of locally advanced or metastatic disease non-amenable to surgery or radiation therapy with curative intent
* At least one measurable lesion >20mm (or >10 mm with spiral CT scan)
* Must have received (and failed) prior treatment with an anthracycline, a taxane, and capecitabine in the adjuvant and/or advanced disease treatment setting
* Women at least 18 years old, with performance status 0-2

Exclusion Criteria:

* Prior treatment with another topoisomerase I inhibitor
* Current enrollment in another clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2003-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of Irinotecan in refractory breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (42):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Anchorage, Alaska
  - Pfizer Investigational Site, Lewistown, Idaho
  - Pfizer Investigational Site, Alton, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Chalmette, Louisiana
  - Pfizer Investigational Site, Covington, Louisiana
  - Pfizer Investigational Site, Mandeville, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Washington, Missouri
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Stony Brook, New York
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Covington, Tennessee
  - Pfizer Investigational Site, Franklin, Tennessee
  - Pfizer Investigational Site, Gallatin, Tennessee
  - Pfizer Investigational Site, Hermitage, Tennessee
  - Pfizer Investigational Site, Lebanon, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Murfreesboro, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, Tyler, Texas
  - Pfizer Investigational Site, Federal Way, Washington
  - Pfizer Investigational Site, Lakewood, Washington
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Vancouver, Washington
  - Pfizer Investigational Site, Yakima, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Argentina (5):
  - Pfizer Investigational Site, Capital Federal, Buenos Aires
  - Pfizer Investigational Site, Córdoba, Córdoba Province
  - Pfizer Investigational Site, Rosario, Santa Fe Province
  - Pfizer Investigational Site, Santa Fe, Santa Fe Province
  - Pfizer Investigational Site, Capital Federal
- Australia (2):
  - Pfizer Investigational Site, South Brisbane, Queensland
  - Pfizer Investigational Site, Frankston, Victoria
- Pfizer Investigational Site, Bogotá, Bogota DC, Colombia
- Pfizer Investigational Site, Wellington, New Zealand

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=CPTAPO-0047-146&StudyName=Irinotecan%20in%20Patients%20with%20Advanced%20Metastatic%20Breast%20Cancer%20Who%20Have%20Experienced%20Failure%20of%20an%20Anthracycline%2C%20a%20Taxane%2C%20and%20C